CLINICAL TRIAL: NCT04361617
Title: A Feasibility Study of Tree Nut and Extra Virgin Olive Oil Supplementation to Improve Cardiometabolic Health
Brief Title: Nuts and Oil Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00065273; UL1TR001420 (NIH)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2021-06

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; extra virgin olive oil; tree nuts; DNA methylation
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Knowledge of intervention arm will not be given to research labs with samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epigenetic age knowledge arm (Active Comparator): Half of the intervention participants will be randomly selected to be informed of epigenetic age before the intervention.
  Interventions: Behavioral: Daily consumption of tree nuts and extra virgin olive oil
- No epigenetic age knowledge arm (Active Comparator): The other half of intervention participants will not be informed of epigenetic age before the intervention.
  Interventions: Behavioral: Daily consumption of tree nuts and extra virgin olive oil

INTERVENTIONS:
Behavioral: Daily consumption of tree nuts and extra virgin olive oil — All participants will receive a 4-week supply of extra virgin olive oil and tree nuts, including unsalted English walnuts, almonds or pistachios (approximately 3-day supply of each type). Participants will be asked to include in their normal diets these products and will be provided recipes and other information that will allow them to replace other foods with the nuts and oil. We will ask participants to consume one ounce of tree nuts per day and two tablespoons of EVOO per day by incorporating these foods into their diet.

SUMMARY:
Metabolic syndrome is considered to be a state of prediabetes and is a major risk factor for cardiovascular disease. Dietary interventions involving extra virgin olive oil (EVOO) supplementation and tree nut consumption can improve cardiometabolic health and reverse metabolic syndrome. The goal of this exploratory study is to establish the feasibility of using a novel measure - epigenetic age - to motivate behavior change and improve cardiometabolic health in individuals with metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a collection of at least three out of five cardiometabolic risk factors including abdominal obesity, hypertension, elevated blood glucose, hypertriglyceridemia, and low high-density lipoprotein cholesterol. MetS is a major risk factor for cardiovascular disease and is considered a state of prediabetes. Improving metabolic parameters through dietary, behavioral, and pharmacological interventions can improve or reverse MetS. For example, increased consumption of extra virgin olive oil (EVOO) and mixed nuts was shown to reduce cardiovascular event rates and reverse MetS in a 5-year study in Spain (PREDIMED study). However, lower levels of adherence to the PREDIMED intervention was found in participants with a higher number of cardiovascular risk factors, larger waist circumference, and lower physical activity levels at baseline. New strategies to convey one's risk of morbidity and mortality at the onset of a dietary intervention may improve intervention adherence, particularly among individuals meeting the criteria for MetS.

A greater DNA methylation-based predicted age relative to chronological age, often referred to as "epigenetic age acceleration", has been associated with many lifestyle factors, including physical activity and diet, as well as components of MetS, including obesity, blood pressure, HDL cholesterol and blood glucose levels.

The investigators hypothesize that the majority of people with MetS have advanced epigenetic aging, and among those that have advanced epigenetic age, learning one's epigenetic age, and epigenetic age-based predicted risk of morbidity and mortality at the onset of a dietary intervention will improve participant adherence to the dietary intervention. Further, the investigators hypothesize that EVOO and tree nut supplementation in participants with MetS and advanced epigenetic age could help reverse MetS and potentially slow epigenetic aging. Therefore, the investigators plan to conduct a feasibility pilot study to:

1. To determine the proportion of participants with MetS with epigenetic age acceleration
2. To assess adherence to daily EVOO and tree nut consumption over a 4-week intervention in participants informed of epigenetic age acceleration at baseline compared to the control group
3. Qualitatively explore how participants perceive epigenetic age, and how participants' experiences would impact the feasibility of a larger clinical intervention in terms of challenges and motivators
4. Compare epigenetic age acceleration before and after the 4-week intervention

For this study the investigators will recruit ~50 individuals with MetS aged 35 years or older. An in-person assessment visit will be scheduled for a morning time and participants will be asked to be fasting and will be instructed to bring their medications to the visit. Candidates will review the informed consent document at an in-person screening with study staff prior to beginning their participation. For all participants providing informed consent, who were fasting and met the MetS criteria at the initial in-person assessment visit, collected blood samples will be used to calculate epigenetic age acceleration. Other measures to be collected include body weight, height, waist circumference, blood pressure, and questionnaires about demographics, health history and health habits. Participants that meet the inclusion criteria during the in-person screening visit will be contacted to schedule a baseline intervention visit.

At the intervention visit, all participants will receive a 4-week supply of EVOO and tree nuts, including unsalted English walnuts, almonds or pistachios (approximately 10-day supply of each type). Participants will be asked to supplement their normal diets with these products and will be provided recipes and other information that will allow them to replace other foods with the nuts and oil. The investigators will ask participants to consume one ounce of tree nuts per day and two tablespoons of EVOO per day by incorporating these foods into their diet. Dietary adherence diaries will be given to measure incorporation of the study foods.

Participants will be randomized to learn about epigenetic age acceleration (arm 1) or not to learn about epigenetic age acceleration (arm 2) in a 1:1 allocation at the baseline visit. Those in the intervention arm 1 that are to learn about epigenetic age acceleration will receive some educational materials and a brief description of epigenetic age acceleration.

A telephone visit will be scheduled to take place at the end of week 1 for additional diet counseling, to assess safety/potential side effects and to collect adherence diaries. A follow-up phone call for compliance assessment and to answer participant questions will be conducted at the end of week 2. A final measurement visit will be scheduled for the end of week 4 for a morning time and participants will be asked to be fasting. At the final measurement visit, the same measures as listed in the in-person assessment visit will be performed and study questionnaires, with the exception of demographics and health history, will be distributed.

After the intervention, participants will be asked to come in for the end of week 4 visit, For participants in the intervention arm 1 (participants educated about epigenetic age acceleration), a self- administered exit questionnaire will be given to qualitatively explore participants' perception of epigenetic age, and challenges and motivators for behavior change during the intervention, The open-ended questions will be designed to ascertain understanding of epigenetic age, and assess the challenges and motivators participants encounter during the intervention.

Participants in both arms will be administered an Intervention Experience Assessment to explore how participant's experiences would impact the feasibility of a larger clinical intervention in terms of challenges and motivators.

This feasibility study, incorporating epigenetic age estimates with a dietary intervention in individuals with MetS, is an initial step in building our understanding of 1) the relationship between MetS and epigenetic age, 2) how epigenetic age estimates may be perceived by patients at high risk for CVD, and 3) will provide preliminary longitudinal data examining the potential to slow epigenetic age acceleration predictions after a 4-week dietary intervention to provide feasibility for a larger future study.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women ≥ 35 years of age
* Metabolic syndrome, defined as > 3 of the following:

Waist circumference >102 cm in men and >88cm in women, triglycerides >150 mg/dL and/or drug treatment for elevated triglycerides, HDL cholesterol <40 mg/dL in men and <50 mg/dL in women and/or drug treatment for reduced HDL cholesterol, systolic blood pressure >130 mm Hg or diastolic blood pressure >85 mmHg and/or antihypertensive drug treatment, and fasting glucose >100 mg/dL or hemoglobin A1c > 5.6% and/or oral hypoglycemic medications.

* Willing to comply with study visits, as outlined in the protocol
* Able to read and speak English
* No allergies or hypersensitivities to olive oil or nuts
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Plans to move from the study area in the next 12 weeks
* Body Mass Index (BMI) > 40 kg/m2
* Dementia that is medically documented or suspected, or clinical evidence of cognitive impairment sufficient to impair protocol adherence
* Candidate with any dietary practice, behavior or attitude that would substantially limit ability to adhere to protocol
* Homebound for medical reasons
* Living in the same household with another participant
* Insulin-dependent Diabetes

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Reynolds, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make IPD available to other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Started | 17 | 17
Completed | 17 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 70 (8) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 11 | 8 | 19
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With MetS With Epigenetic Age Acceleration
Description: To characterize the relationship between MetS and epigenetic aging, we will examine epigenetic age acceleration prevalence among the 50 participants with metabolic syndrome.
Time Frame: In-person 1 day assessment visit
Population: 3 samples failed DNAm QC analyses - 1 sample failed QC analyses
Measure: Number; unit: proportion of participants AgeAccelGrim>
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Number analyzed (Participants) | 14 | 15
proportion of participants AgeAccelGrim> | 0.21 | 0.53

2. Primary Outcome: Proportion of Days for Which EVOO Was Taken
Description: Adherence for each participant will be measured as the proportion of days in 4 weeks for which EVOO was taken
Time Frame: 4 weeks
Population: 3 samples failed DNAm QC analyses - 1 sample failed QC analyses
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Number analyzed (Participants) | 14 | 15
proportion of days | 0.96 (0.08) | 0.97 (0.04)

3. Primary Outcome: Proportion of Days for Which Nuts Were Taken
Description: Adherence for each participant will be measured as the proportion of days in 4 weeks for which nuts were taken
Time Frame: 4 weeks
Population: 3 samples failed DNAm QC analyses - 1 sample failed QC analyses
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Number analyzed (Participants) | 14 | 15
proportion of days | 0.997 (0.010) | 0.997 (0.041)

4. Primary Outcome: Proportion of Days for Which Nuts and EVOO Were Taken
Description: Adherence for each participant will be measured as the proportion of days in 4 weeks for which both nuts and of EVOO were taken
Time Frame: 4 weeks
Population: 3 samples failed to generate DNAm data passing QC analyses 1 sample failed to generate DNAm data passing QC analyses
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Number analyzed (Participants) | 14 | 15
proportion of days | 0.948 (0.076) | 0.967 (0.041)

5. Primary Outcome: Percentage of Participants Would be Able to Continue Eating the Tree Nuts and EVOO for a Study Like This Lasting 3-4 Years
Description: Qualitative interview with open-ended questions designed to ascertain participant understanding of epigenetic age, and assess the challenges and motivators participants encountered during the intervention. Will be assessed using qualitative analysis methods.
Time Frame: After 4-week intervention
Population: % that would be able to continue eating the tree nuts and EVOO for a study like this lasting 3-4 years
Measure: Number; unit: Percentage of Participants
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Number analyzed (Participants) | 17 | 15
Percentage of Participants | 76 | 93

6. Secondary Outcome: Changes in Epigenetic Age Acceleration
Description: The investigators will compare epigenetic age acceleration before and after the 4-week intervention via DNA methylation test.DNA methylation profiles (beta-value, after adjustment chip and position effects) at 1,030 unique DNA methylation profiles will be used for epigenetic age acceleration predictions, using the DNA GrimAge predictor. The investigators will calculate predicted lifespan and regress predicted lifespan on chronological age to produce estimates of epigenetic age acceleration.
Time Frame: In-person 1 day assessment visit vs. final 1 day visit after 4-week intervention
Population: 3 samples failed to generate DNAm data passing QC analyses - 1 sample failed to generate DNAm data passing QC analyses
Measure: Mean (Standard Deviation); unit: AgeAccelGrim (years)
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
Number analyzed (Participants) | 14 | 15
AgeAccelGrim (years) | -0.2 (1.4) | 0.1 (1.3)

ADVERSE EVENTS:
Time Frame: Reporting time frame (ex. Baseline through 4 weeks): Intervention visit through final in person visit
Arm/Group | Epigenetic Age Knowledge Arm | No Epigenetic Age Knowledge Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epigenetic Age Knowledge Arm (N=17) | No Epigenetic Age Knowledge Arm (N=17)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (3) — Nausea
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Hyperglycemia
Pruritus (Infections and infestations) | 1 (1) | 0 (0) — Pruritus
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Hypotension
Weight Gain (Endocrine disorders) | 1 (1) | 0 (0) — Weight Gain
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0) — Indigestion
Upset Stomach (Gastrointestinal disorders) | 2 (2) | 0 (0) — Upset Stomach
bloating or increased bloating (Gastrointestinal disorders) | 1 (5) | 0 (0) — bloating or increased bloating
Increased stool frequency (Gastrointestinal disorders) | 1 (1) | 0 (0) — Increased stool frequency
Loose Bowel movement (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Loose Bowel movement
Gas/Belching (Gastrointestinal disorders) | 1 (3) | 0 (0) — Gas/Belching
Stye in eye (Eye disorders) | 1 (1) | 0 (0) — Stye in eye
Sinus HA with nose bleed (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Sinus HA with nose bleed
Stomach bug with diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Stomach bug with diarrhea
Worsening knee pain and inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Worsening knee pain and inflammation
Lips raw on inside (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Lips raw on inside
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Carpal tunnel
Decreased frequency of bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) — Decreased frequency of bowel movements
Explosive bowel movement) (Gastrointestinal disorders) | 0 (0) | 1 (1) — Explosive bowel movement)
Fatigue (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Fatigue
Infection- Leg sore (Infections and infestations) | 0 (0) | 1 (1) — Infection- Leg sore
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) — Vomiting
Acid reflux/ increased acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) — Acid reflux/ increased acid reflux
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) — Constipation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT04361617/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT04361617/ICF_000.pdf